CLINICAL TRIAL: NCT06444880
Title: Phase II Trial of Ubamatamab Alone or in Combination With Cemiplimab in MUC16-Expressing SMARCB1-Deficient Malignancies
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-1062; NCI-2024-04755 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-05-30; First posted 2024-06-06 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: SMARCB1-Deficient Malignancies
MeSH Terms: interventions — cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Stage I (Experimental): Stage 1 of study treatment involves being given ubamatamab by itself by vein. The first dose will be given over about 4 hours. Depending on how participants respond, later doses may be given over shorter periods of time (possibly down to 30 minutes per infusion). Participants dose of ubamatamab will be increased from a starting dose on Day 1 to a full dose on Day 15.
  Participants will receive ubamatamab 1 time every week for the first 4 weeks, then every 3 weeks after that, unless the disease gets worse or intolerable side effects occur.
  • If the disease gets worse after completing 6 weeks of treatment, participants will move to Stage 2 and receive combination therapy.
  Interventions: Drug: Ubamatamab
- Stage 2 (Experimental): Participants in Stage 2 will begin receiving ubamatamab and cemiplimab.
  * If participants are enrolled directly into Stage 2, but did not have therapy with ubamatamab alone, participants will receive ubamatamab 1 time each week for 4 weeks, before beginning combination therapy.
  * If participants have already completed Stage 1 and are moving on to Stage 2, participants will begin with combination therapy.
  During Stage 2, ubamatamab is given by vein over 30 minutes to 4 hours, as described above. Cemiplimab is given by vein over 30 minutes.
  Interventions: Drug: Ubamatamab; Drug: Cemiplimab

INTERVENTIONS:
Drug: Ubamatamab — Given by IV
Drug: Cemiplimab — Given by IV
  Arms: Stage 2

SUMMARY:
To find out if ubamatamab, given by itself or in combination with cemiplimab, can help to control the disease in participants with renal medullary carcinoma (RMC) and epithelioid sarcoma (ES).

DETAILED DESCRIPTION:
Primary Objectives • To determine the objective response rate (ORR) and disease control rate (DCR), per RECIST 1.1, of ubamatamab alone and in combination with cemiplimab in patients with locally advanced or metastatic MUC16-expressing SMARCB1-deficient malignancies, RMC or ES, who have progressed on at least one prior line of therapy.

Secondary Objectives

• To determine the efficacy and safety of ubamatamab alone or in combination with cemiplimab in participants with locally advanced or metastatic MUC16-expressing SMARCB1-deficient malignancies such as RMC or ES who have progressed on at least one prior line of therapy. Efficacy will be measured by overall survival (OS), progression-free survival (PFS), and duration of response (DOR).

Exploratory Objectives

* To determine the objective response rate (ORR) and disease control rate (DCR), per RECIST 1.1, of the overall strategy of ubamatamab alone followed by combination with cemiplimab in participants with locally advanced or metastatic MUC16-expressing SMARCB1-deficient malignancies, RMC or ES, who have progressed on at least one prior line of therapy.
* To evaluate potential biomarkers, such as serum CA-125 and tumor tissue MUC16 expression levels for participant stratification, and to determine via the molecular profiling of biopsy and blood specimens, the mechanisms of resistance to ubamatamab alone or in combination with cemiplimab.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with locally advanced or metastatic RMC (RMC cohort) or ES (ES cohort) histologically confirmed by expert pathology review and loss of SMARCB1 staining by IHC. Participants with advanced or metastatic unclassified renal cell carcinoma with medullary phenotype (a rare SMARCB1 negative RMC variant occurring in individuals without sickle hemoglobinopathies) are also eligible for the RMC cohort.
2. Eligible participants should either demonstrate serum CA-125 levels ≥ 70 units/ml during screening or positive H score of >25 for MUC16 (CA-125) by IHC in tumor tissues collected within 12 months from screening as noted in participant EMR:

   1. The H score is calculated using the standard formula commonly used in IHC: H score = [(0 x % negative cells) + (1 x % weak positive cells) + (2 x % moderate positive cells) + (3 x % strong positive cells). For instance, if 50% of tumor cells show weak staining, 30% of tumor cells show moderate staining, and 20% of cells show strong staining, the H-score would be: (50×1)+(30×2)+(20×3)=50+60+60=170.
   2. If serum CA-125 ≥ 70 units/ml then participants will be enrolled without delay. IHC for MUC16 will be used as a correlative biomarker but not for trial eligibility.
   3. If serum CA-125 < 70 units/ml then for trial eligibility, MUC16 expression should be checked by IHC in tumor tissues collected within 12 months from screening:

   i. If H score is < 25 then the patient will not be eligible for the trial ii. If H score ≥ 25 then the patient will be eligible for the trial
3. Participants will be eligible in the RMC cohort regardless of whether they have had prior nephrectomy or still have their primary tumor in-situ.
4. Participants must have at least one measurable site of disease, defined as a lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) and measures ≥ 15 mm with conventional techniques or ≥ 10 mm with more sensitive techniques such as MRI or CT scan. If the patient has had previous radiation to the marker lesion(s), there must be evidence of progression since the radiation.
5. Participants must have progressed on at least one line of prior therapy.
6. There must be evidence of progression on or after last treatment regimen received.
7. ECOG performance status 0-1

   a. NOTE: If participant is unable to walk due to paralysis, but is mobile in a wheelchair, participant is considered to be ambulatory for the purpose of assessing their performance status.
8. Age (at the time of consent/assent): ≥ 18 years

   a. RMC is the third most common renal cell carcinoma in children and young adults in the United States21 and while we will initially enroll participants aged ≥18 years old, we will in coordination with Regeneron consider allowing pediatric participants ≥12 years old if no trial limiting toxicities (TOX), as defined in Section 9.1.2., after the interim analysis of the first 10 participants enrolled and based on the accumulated pharmacokinetic / pharmacodynamic data of ubamatamab in this population at that time. If these criteria are fulfilled, then adolescent participants age 12 years and older will be allowed with signed assent and parental consent according to institutional guidelines and requirements, as long as their weight is >40 kg given that this is the lower weight limit for which safety following ubamatamab with or without cemiplimab exposure has been ascertained.
9. Consent to MD Anderson companion laboratory protocol 2014-0938
10. Participants must have adequate organ and marrow function as defined below:

    Hemoglobina ≥ 9 g/dl (treatment allowed) Absolute neutrophil countb ≥ 1,000/µL Platelets ≥ 75,000/µL Total bilirubin ≤ 1.5 mg/dl AST(SGOT) or ALT (SGPT) ≤ 2.5 X institutional ULN, except in known hepatic metastasis, wherein may be ≤ 5 x ULN Serum Creatininec ≤ 1.5 x ULN by gender (as long as patient does not require dialysis)

    a May receive transfusion within the screening period b Without growth factor support (filgrastim or pegfilgrastim) for at least 14 days c If creatinine is not <1.5×ULN, then calculate by Cockcroft-Gault methods or local institutional standard and CrCl must be >30 mL/kg/1.73 m2
11. Participants with controlled brain metastases are allowed on protocol if the brain metastases were surgically resected or treated with radiosurgery or Gamma knife, without recurrence or edema for 1 month (4 weeks). Participants actively requiring glucocorticoids for uncontrolled brain or leptomeningeal metastases are not eligible.
12. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of the study drug.
13. Women must not be breastfeeding.
14. WOCBP must agree to follow instructions for method(s) of contraception from the time of registration for treatment for the duration of treatment with study drug (s) plus 5 half-lives of study drug (s) plus 30 days (duration of ovulatory cycle) for a total of 5 months post treatment completion. Men must agree to effective contraception from the time of registration for treatment to 7 months post last protocol treatment.

    Investigators shall counsel WOCBP and male participants who are sexually active with WOCBP on the importance of pregnancy prevention and the implications of an unexpected pregnancy Investigators shall advise WOCBP and male participants who are sexually active with WOCBP on the use of highly effective methods of contraception. Highly effective methods of contraception have a failure rate of < 1% per year when used consistently and correctly.

    Approved methods of birth control are as follows: Hormonal contraception (i.e. birth control pills, injection, implant, transdermal patch, vaginal ring), Intrauterine device (IUD), Tubal Ligation or hysterectomy, Patient/Partner post vasectomy, Implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.

    Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 7 months after completion of ubamatamab/cemiplimab administration.

    The effects of ubamatamab/cemiplimab on the developing human fetus are unknown. For this reason and because immunotherapy agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. (Refer to Pregnancy Assessment Policy MD Anderson Institutional Policy # CLN1114). This includes all female participants, between the onset of menses (as early as 8 years of age) and 55 years unless the patient presents with an applicable exclusionary factor which may be one of the following:
    * Postmenopausal (no menses in greater than or equal to 12 consecutive months).
    * History of hysterectomy or bilateral salpingo-oophorectomy.
    * Ovarian failure (Follicle Stimulating Hormone and Estradiol in menopausal range, who have received Whole Pelvic Radiation Therapy).
    * History of bilateral tubal ligation or another surgical sterilization procedure.
15. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Participants must not have any other malignancies within the past 2 years except for in situ carcinoma of any site, or adequately treated (without recurrence post-resection or post-radiotherapy) carcinoma of the cervix or basal or squamous cell carcinomas of the skin, ductal carcinoma in situ of the breast or low-risk early stage prostate adenocarcinoma with negligible risk of metastasis or death
2. Participants previously treated with T-cell-redirecting bispecific antibodies or MUC16-targeted therapies (including vaccines) are excluded. Participants who received CAR-T therapies within 30 days of first dose of study drug are also excluded. However, participants previously treated with immune checkpoint therapies such as anti-PD1, anti-PD-L1, anti-CTLA-4, or anti-LAG-3 immune checkpoint inhibitors are eligible, as long as they have been off these therapies for at least 60 days (~3 half-lives) prior to initiation of study treatment with ubamatamab.
3. Participants currently receiving anticancer therapies or who have received anticancer therapies (including chemotherapy and targeted therapies such as tazemetostat) within 2 weeks (14 days) prior to study Day 1 are excluded. Participants who have completed palliative radiation therapy more than 14 days prior to the first dose of the combination immunotherapy are eligible.
4. Participants with persistent grade ≥2 adverse events from prior systemic therapies that would confound timely detection of immune-related adverse events due to ubamatamab and/or cemiplimab or otherwise hinder patient participation in the clinical trial.
5. Participants, who have had a major surgery or significant traumatic injury (injury requiring > 4 weeks (28 days) to heal) within 4 weeks (28 days) of start of study drug, participants who have not recovered from the side effects of any major surgery (defined as requiring general anesthesia).
6. Participants who have organ allografts.
7. Known or suspected autoimmune disease. Participants with a history of inflammatory bowel disease (including Crohn's disease and ulcerative colitis) and autoimmune disorders such as rheumatoid arthritis, systemic progressive sclerosis [scleroderma], Systemic Lupus Erythematosus or autoimmune vasculitis [e.g., Wegener's Granulomatosis] are excluded from this study. Participants with a history of Hashimoto's thyroiditis only requiring hormone replacement, Type I diabetes, or psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are allowed to participate.
8. Uncontrolled infection with human immunodeficiency virus, hepatitis B or hepatitis C infection; or diagnosis of immunodeficiency.

   1. Participants with HIV who have controlled infection (undetectable viral load with the exception of clinically insignificant blips and CD4 count above 350 either spontaneously or on a stable antiviral regimen) are permitted.
   2. Participants with hepatitis B surface antigen positive (HepBsAg+) who have controlled infection (serum hepatitis B virus DNA PCR that is below the limit of detection AND receiving antiviral therapy for hepatitis B) are permitted.
   3. Participants with HBsAg negative but total HBV core antibody positive (HBc Ab+) are permitted with the following requirements: Serum HBV DNA PCR should be tested and if it is above the limit of detection at screening then antiviral therapy for HBV must be initiated prior to study entry. If serum HBV DNA PCR is below the limit of detection periodic monitoring of HBsAg must be performed every 12 months +/- 3 months.
   4. Participants who are Hepatitis C virus antibody positive (HCV Ab +) who have controlled infection (undetectable HCV RNA by PCR either spontaneously or in response to a successful prior course of anti-HCV therapy) are permitted.
9. Any underlying medical condition, which in the opinion of the Investigator, will make the administration of study drug hazardous or obscure the interpretation of adverse events, such as a condition associated with frequent diarrhea, uncontrolled nausea or vomiting. Patients with active COVID-19 disease as indicated by a positive polymerase reaction (PCR) test are excluded. Participants with previous COVID-19 disease are allowed if ≥30 days from last positive test, and COVID-19 symptoms have resolved and/or PCR test is now negative.
10. Participants must not be scheduled to receive another experimental drug while on this study.
11. Participants who are on high dose steroid (e.g., > 10mg prednisone daily or equivalent) or other more potent immune suppression medications (e.g., infliximab). Topical, inhaled, intra-articular, ocular, or intranasal corticosteroids (with minimal systemic absorption) are allowed. A brief course (<48 hours) of systemic corticosteroids for prophylaxis (eg, from contrast dye allergy) is permitted. Physiological corticosteroid replacement therapy for adrenal insufficiency (up to hydrocortisone 30 mg / daily or equivalent) is also permitted.
12. Left ventricular ejection fraction (LVEF) assessment with documented LVEF < 50% by transthoracic echocardiogram (TTE) within 6 months prior to start of study treatment. In cases of LVEF 45-50% in absence of clinical symptoms, after review and clearance by cardiologist, the patient may be enrolled.
13. Active myocarditis, regardless of etiology.
14. Moderate to large pericardial effusion (eg, > approximately 100 mL) as measured by echocardiogram at baseline. Multigated acquisition (MUGA) is not sufficient for evaluating pericardial effusion.
15. Has a history of any clinically significant arrhythmia including atrial fibrillation or implantation of a pacemaker or defibrillator.
16. Participants who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:

    1. Symptomatic congestive heart failure of New York heart Association Class III or IV
    2. Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months of start of study drug, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease
    3. Systemic fungal, bacterial, viral, or other infection that is not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement) despite appropriate antibiotics or other treatment.
    4. Participants with a history of major psychiatric illness judged unable to fully understand the investigational nature of the study and the risks associated with the therapy.
17. Participants must not have history of other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of ubamatamab or cemiplimab or that might affect the interpretation of the results of the study or render the participant at high risk from treatment complications.
18. Participants should not receive immunization with attenuated live vaccines within 30 days of planned start of study medication.

    a. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
19. Female participants who are pregnant or breast feeding, or adults of reproductive potential who are not willing to use effective birth control methods as defined above.
20. Any participants who cannot be compliant with the appointments required in this protocol must not be enrolled in this study.
21. History of allergic reactions attributed to compounds of similar chemical or biologic composition to ubamatamab or cemiplimab.
22. Participants with psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year.
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Pavlos Msaouel, MD,PHD,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Connolly DM, Revon-Riviere G, Chami R, Mills D, Coblentz AC, Uldrick TS, Knorr DA, Goncalves P, Dobosz M, Jalal S, Cohen-Gogo S, Morgenstern DA. Mucin 16-Directed Therapy in Pediatric Sarcomas: Case Evidence of Ubamatamab Efficacy in Epithelioid Sarcoma and Its Implications for Other Sarcoma Subtypes. JCO Precis Oncol. 2025 Aug;9:e2500404. doi: 10.1200/PO-25-00404. Epub 2025 Aug 1. PMID 40749151
- See also: MD Anderson Cancer Center — http://www.mdanderson.org